CLINICAL TRIAL: NCT03594331
Title: A Phase I, First-in-Human Single Center Study in Healthy Adult Volunteers to Assess the Gastric Gluten-Degradation Activity of PvP001
Brief Title: Gastric Gluten-Degradation Activity of PvP001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding stopped
Sponsor: Danielle Kim Turgeon (Other)
Collaborators: PvP Biologics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00122254
Record Dates: First submitted 2018-06-21; First posted 2018-07-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Digestive System Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gluten Exposure Group 1 (Experimental): This group will ingest the drug and then consume a study meal containing a low level of gluten. In four separate visits, each subject will be administered low-dose PvP001, medium-dose PvP001, high-dose PvP001 and placebo, with blinding to the dose of PvP001 and to which visit placebo is given.
  Interventions: Drug: Low-dose PvP001; Drug: Medium-dose PvP001; Drug: High-dose PvP001; Drug: Placebo
- Gluten Exposure Group 2 (Experimental): This group will ingest the drug and then consume a study meal containing a medium level of gluten. In four separate visits, each subject will be administered low-dose PvP001, medium-dose PvP001, high-dose PvP001 and placebo, to the dose of PvP001 and to which visit placebo is given.
  Interventions: Drug: Low-dose PvP001; Drug: Medium-dose PvP001; Drug: High-dose PvP001; Drug: Placebo
- Gluten Exposure Group 3 (Experimental): This group will ingest the drug and then consume a study meal containing a high level of gluten. In four separate visits, each subject will be administered low-dose PvP001, medium-dose PvP001, high-dose PvP001 and placebo, with blinding to the dose of PvP001 and to which visit placebo is given.
  Interventions: Drug: Low-dose PvP001; Drug: Medium-dose PvP001; Drug: High-dose PvP001; Drug: Placebo

INTERVENTIONS:
Drug: Low-dose PvP001 — Low-dose PvP001
Drug: Medium-dose PvP001 — Medium-dose PvP001
Drug: High-dose PvP001 — High-dose PvP001
Drug: Placebo — 100 mL liquid with no drug

SUMMARY:
This is a single blind, dose escalating, placebo-controlled, crossover study of gluten-degrading drug PvP001 administered to healthy volunteers (age 18-64 years). Subjects will be randomized to one of three groups representing different levels of gluten exposure - low, medium, or high - in a single meal. Within each gluten exposure group, increasing doses of PvP001 (or placebo) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* Able to maintain a gluten-free diet (GFD) for 24 hours prior to each of visits 1-4;
* Able to abstain from alcohol consumption 72 hours before and 72 hours after each visit;
* Able to tolerate the placement, presence, and manipulation of an oro-gastro-duodenal (OGD) tube;
* Women of child-bearing potential and men whose partners are women of child-bearing potential must be willing to use acceptable birth control for the duration of the study;
* Able to read and understand English;
* Able to provide written informed consent

Exclusion Criteria:

* Any condition or abnormality, current or past, that, in the opinion of the investigator, would compromise the safety of the subject, or would interfere with or complicate study procedures or assessments.
* No current or recent (within 14 days prior to each study visit, clinical laboratory testing, and ECG) use of over-the-counter or prescription medications via any route of administration, except for oral contraceptives for birth control (provided they have been used regularly for at least the past 3 months). Other medications used regularly at stable doses may be acceptable at the discretion of the study doctor.
* Current symptoms of congestion, upper respiratory tract infection, or acute illness
* Chronic viral infection or immunodeficiency condition
* Any female who is pregnant, planning to become pregnant during the study, or breast-feeding
* History of intolerance, hypersensitivity, or reaction to wheat or other grains, gluten, or any other food or food ingredient (including an additive or preservative) in the study meal;
* Receipt of an investigational medication within four weeks prior to the screening visit or from the screening visit through the final visit;
* Alcohol consumption >5 drinks/week or any alcohol consumption within the 72 hours prior to each study exposure visit or a positive breathalyzer test result at any study visit;
* Illicit or recreational drug use in the past 12 months or positive urine drug screen at the screening visit;
* History of smoking, nicotine, or tobacco use in the past 12 months;
* History or high risk of noncompliance with treatment or visits.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | 2 weeks from each exposure.
  The number of treatment emergent adverse events at each dosage level
Percentage of treatment emergent adverse events | 2 weeks from each exposure.
  The percentage of treatment emergent adverse events at each dosage level
Side effects of study drug | 12 months
  Side effects are assessed by the PI using a 5-scale, 9-question Gastrointestinal Symptoms Questionnaire (GSQ) to be self-administered by the subject at 16 time-points throughout the five-visit (including screening) study. Each of the 9 questions will be given a numerical score (0-4 where 0 is none and 4 is very severe) and compared to baseline score and placebo scores any increase of >1 point over the average baseline and placebo score will be considered an AE and graded based on the severity reported.
Efficacy as measured by the lowest dose to degrade highest amount of gluten | 12 months
  The lowest dose of PvP001 that degrades the highest amount of gluten in a standardized study meal

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States